CLINICAL TRIAL: NCT05391880
Title: A Randomized, Double-Blind, Placebo-Controlled Study of Orally Administered BEBT-503 to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single Ascending Doses (SAD) and Multiple Ascending Doses (MAD) in Healthy Subjects
Brief Title: Study of Orally Administered BEBT-503 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BeBetter Med Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GBMT-503-P01
Record Dates: First submitted 2022-05-12; First posted 2022-05-26 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2022-05

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug:BEBT-503 (Experimental): BEBT-503
  Interventions: Drug: BEBT-503 20mg; Drug: BEBT-503 40mg; Drug: BEBT-503 80mg; Drug: BEBT-503 120mg; Drug: BEBT-503 180mg
- Drug: Placebo (Placebo Comparator): Placebo
  Interventions: Drug: placebo 20mg; Drug: placebo 40mg; Drug: placebo 80mg; Drug: placebo 120mg; Drug: placebo 180mg

INTERVENTIONS:
Drug: BEBT-503 20mg — BEBT-503 capsule
  Arms: Drug:BEBT-503
Drug: BEBT-503 40mg — BEBT-503 capsule
  Arms: Drug:BEBT-503
Drug: BEBT-503 80mg — BEBT-503 capsule
  Arms: Drug:BEBT-503
Drug: BEBT-503 120mg — BEBT-503 capsule
  Arms: Drug:BEBT-503
Drug: BEBT-503 180mg — BEBT-503 capsule
  Arms: Drug:BEBT-503
Drug: placebo 20mg — placebo capsule
  Arms: Drug: Placebo
Drug: placebo 40mg — placebo capsule
  Arms: Drug: Placebo
Drug: placebo 80mg — placebo capsule
  Arms: Drug: Placebo
Drug: placebo 120mg — placebo capsule
  Arms: Drug: Placebo
Drug: placebo 180mg — placebo capsule
  Arms: Drug: Placebo

SUMMARY:
This is a Phase I, randomized, double-blind, placebo-controlled, first-in-human study in which the safety, tolerability, and pharmacokinetic of orally administered BEBT-503 will be assessed in healthy adult subjects.

The study will consist of 2 parts: a SAD phase (Part A) enrolling a total of 5 cohorts of healthy subjects; a MAD phase (Part B) enrolling 2 cohorts of healthy subjects; One cohort of Part A will receive BEBT-503 under both fasted and fed conditions to investigate the effect of food

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, of any race, between 18 and 55 years of age, inclusive.
2. Body mass index (BMI) of 18.0 to 30.0 kg/m2 (inclusive) with a minimum body weight of 50 kg. Participants with a BMI up to 32.0 kg/m2 may be enrolled with the sponsor's approval
3. In good health, determined by no clinically significant findings from medical history, physical examination, 12-lead ECG, vital signs measurements, and clinical laboratory evaluations (congenital nonhemolytic hyperbilirubinemia, eg, suspicion of Gilbert's syndrome based on total and direct bilirubin, is not acceptable) at Screening and Check-in as assessed by the Investigator (or designee), as applicable.
4. Resting heart rate ≥ 45 bpm and ≤ 90 bpm with a single 12-lead ECG at Screening.
5. Females will not be pregnant or lactating, and females of childbearing potential and males will agree to use contraception.
6. Male subjects must agree to refrain from sperm donation and females should refrain from ova donation from the date of Check-in (Day-1) until 90 days after the Follow-up visit.
7. Participants have ability to swallow and retain oral medication.
8. Able to comprehend and willing to sign an Information and Consent Form and to abide by the study restrictions.

Exclusion Criteria:

1. Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the Investigator (or designee).
2. History of febrile illness within 7 days prior to the first dose of study drug or subjects with evidence of active infection.
3. History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator (or designee).
4. History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs (uncomplicated appendectomy and hernia repair will be allowed, but not cholecystectomy).
5. History of malignancy (cured basal cell or squamous cell carcinoma of the skin, ductal carcinoma in situ are eligible).
6. Presence of a malabsorption syndrome possibly affecting drug absorption (eg, Crohn's disease or chronic pancreatitis).
7. Any of the following:

   1. corrected QT interval by Fridericia formula> 450 msec confirmed by repeat measurement.
   2. QRS duration > 120 msec confirmed by repeat measurement.
   3. PR interval > 220 msec confirmed by repeat measurement.
   4. findings which would make corrected QT interval measurements difficult or corrected QT interval data uninterpretable.
   5. history of additional risk factors for torsade de pointes (eg, heart failure, hypokalemia, family history of long QT syndrome).
8. History of alcoholism or drug/chemical abuse within 6 months prior to Check-in.
9. Alcohol consumption of > 21 units per week for males and > 14 units per week for females. One unit of alcohol equals ½ pint (285 mL) of beer or lager, 1 glass (125 mL) of wine, or 1/6 gill (25 mL) of spirits.
10. Positive alcohol breath test result or positive urine drug screen (confirmed by repeat) at Screening or Check-in.
11. Positive hepatitis panel and/or positive human immunodeficiency virus (HIV) test.
12. Participation in a clinical study involving administration of an investigational agent or vaccine (new chemical entity) or having received a biological product in the past 90 days prior to dosing.
13. Use or intend to use any medications/products known to alter drug absorption, metabolism, or elimination processes, including St. John's wort, within 30 days prior to dosing, unless deemed acceptable by the Investigator (or designee).
14. Use or intend to use any prescription medications/products other than hormone replacement therapy, oral, implantable, transdermal, injectable, or intrauterine contraceptives within 14 days prior to dosing, unless deemed acceptable by the Investigator (or designee).
15. Use or intend to use slow-release medications/products considered to still be active within 14 days prior to Check-in, unless deemed acceptable by the Investigator (or designee).
16. Use or intend to use any nonprescription medications/products including vitamins, minerals, and phytotherapeutic/herbal/plant-derived preparations within 7 days prior to Check-in, unless deemed acceptable by the Investigator (or designee).
17. Use of tobacco- or nicotine-containing products within 1 month prior to Check-in, or positive cotinine at Screening or Check-in.
18. Receipt of blood products within 2 months prior to Check-in and donation of blood from 3 months prior to Screening, plasma from 2 weeks prior to Screening, or platelets from 6 weeks prior to Screening.
19. Any major surgery within 4 weeks prior to first dosing.
20. Poor peripheral venous access.
21. Have previously completed or withdrawn from this study investigating BEBT-503, and have previously received the investigational product.
22. Subject who, in the opinion of the Investigator (or designee), should not participate in this study.
23. Subject is not willing to minimize or avoid exposure to natural or artificial sunlight (tanning beds or ultraviolet A/B treatment) following administration of study drug until 24 hours after the last dose.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2022-08-26 (Actual); Primary Completion 2023-05-29 (Actual); Study Completion 2023-07-05 (Actual)

PRIMARY OUTCOMES:
single dose safety | from baseline to Day10
  Number of the Adverse Events that are related to the single dose treatment from baseline to Day 10
multiple dose safety | from baseline to Day18
  Number of the Adverse Events that are related to the multiple dose treatment from baseline to Day 18

SECONDARY OUTCOMES:
AUC0-∞ after single dose | Pre-dose to 48 hours postdose
  PK characteristics after single dose
Cmax after single dose | Pre-dose to 48 hours postdose
  PK characteristics after single dose
t1/2 after single dose | Pre-dose to 48 hours postdose
  PK characteristics after single dose
Tmax after single dose | Pre-dose to 48 hours postdose
  PK characteristics after single dose
CL/F after single dose | Pre-dose to 48 hours postdose
  PK characteristics after single dose
Vz/F after single dose | Pre-dose to 48 hours postdose
  PK characteristics after single dose
AUC0-τ after multiple dose | Day 1: pre-am dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, and 24hours post-am dose Days 4 to 9: pre-am dose Day 10: pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16 and 24 hours post-final dose
  PK characteristics after multiple dose
AUC0-∞ after multiple dose | Day 1: pre-am dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, and 24hours post-am dose Days 4 to 9: pre-am dose Day 10: pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16 and 24 hours post-final dose
  PK characteristics after multiple dose
Cmax after multiple dose | Day 1: pre-am dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, and 24hours post-am dose Days 4 to 9: pre-am dose Day 10: pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16 and 24 hours post-final dose
  PK characteristics after multiple dose
t1/2 after multiple dose | Day 1: pre-am dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, and 24hours post-am dose Days 4 to 9: pre-am dose Day 10: pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16 and 24 hours post-final dose
  PK characteristics after multiple dose
Tmax after multiple dose | Day 1: pre-am dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, and 24hours post-am dose Days 4 to 9: pre-am dose Day 10: pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16 and 24 hours post-final dose
  PK characteristics after multiple dose
Cmin after multiple dose | Day 1: pre-am dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, and 24hours post-am dose Days 4 to 9: pre-am dose Day 10: pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16 and 24 hours post-final dose
  PK characteristics after multiple dose
RAAUC0-τ after multiple dose | Day 1: pre-am dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, and 24hours post-am dose Days 4 to 9: pre-am dose Day 10: pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16 and 24 hours post-final dose
  PK characteristics after multiple dose
RACmax after multiple dose | Day 1: pre-am dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, and 24hours post-am dose Days 4 to 9: pre-am dose Day 10: pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16 and 24 hours post-final dose
  PK characteristics after multiple dose
effect of food on the single oral dose AUC0-∞ | Pre-dose to 48 hours postdose
  effect of food on the single oral dose PK
effect of food on the single oral dose Cmax | Pre-dose to 48 hours postdose
  effect of food on the single oral dose PK
effect of food on the single oral dose Tmax | Pre-dose to 48 hours postdose
  effect of food on the single oral dose PK
effect of food on the single oral dose t1/2 | Pre-dose to 48 hours postdose
  effect of food on the single oral dose PK
effect of food on the single oral dose CL/F | Pre-dose to 48 hours postdose
  effect of food on the single oral dose PK
effect of food on the single oral dose Vz/F | Pre-dose to 48 hours postdose
  effect of food on the single oral dose PK
metabolites of BEBT-503 in urine | Pre-dose to 48 hours postdose
  metabolites analysis
metabolites of BEBT-503 in plasma | Pre-dose to 48 hours postdose
  metabolites analysis

CONTACTS AND LOCATIONS:
Overall Officials: Jason Lickliter, CMO, Study Director — Nucleus Network
Locations (1):
- Nucleus Network Pty Ltd, Melbourne, Australia